CLINICAL TRIAL: NCT05362448
Title: Assessment of Cerebellar Ataxia Associated With Ventral Intermediate Median Nucleus Deep Brain Stimulation in Essential Tremor: a Multimodal Neurophysiologic Study
Brief Title: Neurophysiologic Assessment of ET Patients Treated by Vim DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Thomas Wirth, Clinical Research Fellow, University College London Hospitals
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 274481
Record Dates: First submitted 2022-04-11; First posted 2022-05-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Essential Tremor
Keywords: Deep brain Stimulation; Ventral Intermediate nucleus; Gait motion analysis; Balance against force perturbation analysis; Computerized spiral test analysis; Frequency
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 80 Hz (Active Comparator): Stimulation with a frequency of 80 Hz
  Interventions: Device: Frequency
- 130 Hz (Active Comparator): Stimulation with a frequency of 130 Hz
  Interventions: Device: Frequency
- 180 Hz (Active Comparator): Stimulation with a frequency of 180 Hz
  Interventions: Device: Frequency
- DBS off (Sham Comparator): Absence of stimulation
  Interventions: Device: Frequency

INTERVENTIONS:
Device: Frequency — First, we will calculate for each patient and each frequency the amplitude therapeutic window (difference between therapeutic and side effect threshold). We will determine an optimal amplitude for each frequency that we will apply in the second part of the study.

SUMMARY:
Essential tremor is a chronic and progressive neurological disease characterized by upper limb tremor. This is one of the most frequent movement disorders. Most of the time the disease worsens over the time, affecting patients' work abilities and in the most severe cases activities of daily living such as eating or dressing. For the most disabled patients, Deep brain stimulation (DBS) of the thalamic ventral intermediate median nucleus (Vim), a procedure consisting in an electrode implantation in a structure of the brain involved in tremor genesis, is the gold standard treatment. While this therapy is most of the time highly effective in alleviating the tremor, some subjects may exhibit gait impairment or upper limb coordination troubles years after the surgery, which are thought to be due to the involuntary stimulation of efferent cerebellar fiber tract. Unfortunately, this DBS induced side effect cannot be systematically avoided and may limit the possibilities of settings adaptation required to control the tremor. Surprisingly, while it could be a valuable therapeutic option for these patients suffering from DBS induced balance troubles, little is known about the effect of varying the rate of stimulation on the gait disorders associated with essential tremor and Vim DBS. The aim of or study is consequently to assess the effect of different frequency of stimulation on tremor, gait and balance disorders as well as on eye movements in patients uni or bilaterally stimulated in the Vim for a severe and medically intractable essential tremor. Patients followed at the National Hospital for Neurology and Neurosurgery (University College London Hospital) will be included. To better characterize the different symptoms, the investigators will use ataxia and tremor rating scale together with 3D gait motion analysis, oculography and computerized spiral test analysis. Our findings might lead to a better understanding of Vim-DBS associated gait disorders in essential tremor.

DETAILED DESCRIPTION:
Essential tremor (ET) is a chronic, progressive neurological disease characterized by a symmetrical 4-12 Hz kinetic tremor constantly affecting hands and arms. The tremor can also involve the neck, the lower limb, the voice, the mouth, the tongue or other body regions. ET is among the most frequent movement disorders, with an estimated prevalence of 0,9% of the global population. While the tremor can be mildly disabling at the beginning of the disease, most patients experience a worsening of their tremor over the time. Eventually, disease progression can lead to severe disability, impacting patients' working abilities and in the most severe cases, activity of daily living. Though ET being a frequent debilitating condition, there are still few therapeutic options for the most disabled patients. Several surgical procedures have been evaluated in ET including Deep brain Stimulation (DBS) of Thalamic Ventral intermediate nucleus (Vim) or within the posterior subthalamic area, surgical thalamotomy, Gamma knife or, more recently, MRI guided focused ultrasound thalamotomy. While Gamma knife and focused ultrasound thalamotomy may be safer due to the absence of craniotomy, Vim-DBS remains currently the reference treatment and the most used procedure for medically refractory ET.

Besides the early side effects of Vim-DBS such as haemorrhagic, ischemic and infectious complications occurring immediately after the electrodes implantation procedure, late side-effects such as cerebellar symptoms including gait or upper limb cerebellar ataxia, paraesthesia, dysarthria, dysphagia, and cognitive difficulties are quite frequent. These long-term consequences of the stimulation may dramatically impact the quality of life of patients suffering from ET years after the surgery and mitigate the benefits of this intervention. Considering gait ataxia, it has been reported that this complication may affect up to 37% of ET patients following Vim-DBS surgery and seem to occur more frequently in patient who had pre-operative gait impairment, greater disease severity, older age and when DBS was performed bilaterally. Upper limb ataxia is also common and characterized by the occurrence or the paradoxical worsening of an intention tremor together with asynergy, dyschronometria and dysdiadochokinesia. It has been shown that this latter can be induced by suprathreshold stimulation.

One of the major assets of Vim-DBS over surgical thalamotomy remain its ability to steadily adapt the current delivered by the electrodes by changing the stimulation parameters. Using traditional Implantable Pulse Generator (IPG), it is possible to modify the stimulation mode (monopolar or bipolar stimulation), amplitude, frequency and pulse width as well as to modify the contacts of the electrodes delivering the current. However, despite DBS being a treatment largely available worldwide as well as being part of the routine care for medically refractory tremor, only few studies have assessed the effects of varying DBS settings on cerebellar symptoms presented by patients suffering from ET and stimulated within the Vim. It has been reported that tremor responds best to amplitude, which is usually increased until a complete resolution of the tremor is obtained. Increasing the stimulation pulse width produces a similar clinical effect and may help to alleviate tremor. Interestingly, it has recently been shown that decreasing the pulse width may improve the gait disorders, widen the therapeutic window and diminishes DBS induced side effects. This clinical finding is supported by the recent dissection of the neuronal network underlying Vim DBS clinical response which suggest that tremor suppression could be due to dentato-rubro-thalamic tract stimulation while gait and limb ataxia could be promoted by the stimulation of the cerebello-rubro-spinal and the rubro-olivo-cerebellar tract meaning the possibility of correcting these side effects by accurately optimizing the DBS parameters.

Among the clinical effect of the different types of parameters, the stimulation frequency has certainly been the less extensively studied in ET. This is at first sight quite surprising given that decreasing the frequency of stimulation of the Subthalamic nucleus (STN) is a valuable therapeutic option in Parkinson's disease especially for patient presenting with dopa-refractory symptoms such as freezing of gait or speech impairment. Lower frequency stimulation has also shown to be beneficial for some patients suffering from dystonia, and it has been suggested that this sustained clinical improvement was obtained by avoiding the stimulation of the structure responsible of side effects.

In comparison, a very low number of studies has focused on the consequences of lower frequency stimulation on tremor. Noteworthy is the fact that most of them have pointed that the tremor suppression was better achieved for a frequency around 100 Hz, with little evidence for a small additional therapeutic effect for frequencies above 130 Hz. Conversely, frequency of 50 Hz or lower seems to not suppress tremor and could even worsen it or induce myoclonic jerks. Based on these clinical findings, it is currently admitted initiating the stimulation with a frequency of 130 Hz and increasing it up to 180 Hz if the therapeutic effect on tremor remains unsatisfying despite concomitant high amplitude and large pulse width. A recent small case series has interestingly shown that some patients presenting with balance disorder years after Vim DBS surgery were having their trouble improved when the stimulation frequency was decreased to 130 Hz. Additionally, there are some evidence that, similarly to short pulse width stimulation, decreasing the frequency up to 100 Hz may help to optimize postural or intention tremor and DBS side effects control by widening the therapeutic window. Taken together, these findings suggest that, similarly to shorter pulse width, a lower frequency of stimulation could be an interesting therapeutic approach for ET patients suffering from balance disorders or upper limb ataxia promoted by Vim-DBS. However, since all the above-mentioned studies were unblinded and non-randomized, the level of evidence supporting such a strategy remain weak. Additionally, none of these works has aimed at evaluating the effect of decreasing DBS frequency on gait and balance, neither by using clinical testing, nor by using quantitative measurement such as 3D motion analysis or computerized posture assessment.

For these reasons, the aim of the present study will be to study the effect of varying Vim-DBS frequency on cerebellar features including gait and upper limb ataxia in ET by using non-invasive quantitative physiological tools, namely computerized spiral test analysis, 3D infrared gait motion analysis, balance measure against force perturbation analysis and oculography.

Patients presenting an ET treated by Vim-DBS stimulation for more than 3 months, followed at the National Hospital of Neurology and Neurosurgery, University College London Hospital, London, United Kingdom will be included.

Regarding the procedure, the investigators will first assess the therapeutic window by estimating the therapeutic and side effect thresholds for three different frequencies (80 Hz-130 Hz-180 Hz). Additionally, the investigators will subsequently analyse balance and gait using a 3D motion analysis system, the tremor using a tablet coupled to a computerized spiral analysis software and eye movements using oculography for the three different settings and with the DBS turned off.

Eventually, the investigators will localize the position of the electrodes and model Volume of Tissue Activated using the DBS planning software Guide-XT® and the pre and postoperative brain MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. No gender specification
3. Patient suffering from severe medically intractable essential tremor and treated by Vim-DBS
4. Willing and able to provide written informed consent

Exclusion Criteria:

1. Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within the last 3 months before study enrolment
2. Patients presenting with other cause(s) of balance or gait disorders (stroke, concomitant neurological, rheumatological or orthopaedic disease, severe hypopallesthesia, visual impairment, neuromuscular or vestibular disorders)
3. Recently implanted patients (<3 months)
4. Patients unable to provide written informed consent (patients presenting with psychiatric or cognitive disorders)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Center of Pressure Displacement | 1 day
  Quantitative continuous variable assessed using balance against force perturbation analysis under the three different DBS settings conditions and with the DBS switched off

SECONDARY OUTCOMES:
Side effect threshold | 1 day
  Amplitude of DBS stimulation needed to induce side effects under the three DBS settings conditions
Therapeutic threshold | 1 day
  Amplitude of DBS stimulation needed to correct tremor under the three DBS settings conditions
Therapeutic window | 1 day
  Difference between side effect threshold and therapeutic threshold under the three DBS settings conditions
Total Energy Delivered | 1 day
  Energy delivered by the pulse generator under the three different DBS settings conditions
Charge density | 1 day
  Charge delivered by the pulse generator under the three different DBS settings conditions
Scale for the Assessment and Rating of Ataxia score | 1 day
  Scoring of cerebellar ataxia under the three different DBS settings conditions and with the DBS switched off
Tremor rating scale score | 1 day
  Scoring of tremor severity under the three different DBS settings conditions and with the DBS switched off
Volume of Tissue Activated | 1 day
  Prediction through imaging of the volume of tissue activated by stimulation under the three different DBS settings conditions
Computerized spiral test analysis (SWVI) | 1 day
  Comparison of spiral width variability index (SWVI) between the four different conditions
Computerized spiral test analysis (AUC) | 1 day
  Comparison of the Area under the curve (AUC) of the acceleration after Fast Fourier Transform between the four different conditions
Computerized spiral test analysis (tremor frequency) | 1 day
  Comparison of the tremor frequency between the four different conditions
Balance motion analysis (CoP initial position) | 1 day
  Comparison of the center of pressure (CoP) initial position and the resisting force between the four different conditions
Balance motion analysis (resisting force) | 1 day
  Comparison of the resisting force between the four different conditions
Gait motion analysis (step length) | 1 day
  Comparison of step length between the four different conditions
Gait motion analysis (number of steps) | 1 day
  Comparison of the number of steps between the four different conditions
Gait motion analysis (stride length) | 1 day
  Comparison of the stride length between the four different conditions
Gait motion analysis (stride velocity) | 1 day
  Comparison of the stride velocity between the four different conditions
Gait motion analysis (normalized double support time) | 1 day
  Comparison of the normalized double support time between the four different conditions
Gait motion analysis (step length asymmetry) | 1 day
  Comparison of the step length asymmetry between the four different conditions
Oculography (fixation index) | 1 day
  Comparison of the fixation index between the four different conditions using eye tracking system
Oculography (saccades velocity) | 1 day
  Comparison of saccades velocity between the four different conditions using eye tracking system
Oculography (saccades latency) | 1 day
  Comparison of saccades latency (ms) between the four different conditions using eye tracking system
Oculography (saccades accuracy index) | 1 day
  Comparison of saccades accuracy index between the four different conditions using eye tracking system
Oculography (VOR gain) | 1 day
  Comparison of the vestibulo-ocular reflex gain (VOR) between the four different conditions using eye tracking system

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No